CLINICAL TRIAL: NCT01010867
Title: A Limited Institution Pilot Trial Evaluating the Safety of Administering the Probiotic, Lactobacillus Plantarum, to Children and Adolescents Undergoing Allogenic Hematopoietic Stem Cell Transplantation (HSCT) - A Pilot Study
Brief Title: Probiotic Use in Children Undergoing Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other); Nemours Children's Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAE0846
Record Dates: First submitted 2009-11-06; First posted 2009-11-10 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Hematopoietic Organs; Disorder
Keywords: Probiotics; Hematopoietic Stem Cell Transplantation; Pediatrics
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lactobacillus plantarum (Experimental): There is a single intervention arm in this study. Target accrual for the intervention is 30 subjects. Subjects receive supplementation with Lactobacillus plantarum strains 299 and 299v.
  Interventions: Drug: Lactobacillus plantarum strains 299 and 299v

INTERVENTIONS:
Drug: Lactobacillus plantarum strains 299 and 299v — Patients will receive a daily dose of Lactobacillus plantarum: 1 x10^8 CFU/kg/day. This supplement will be supplied in sachets of powder and will be mixed in water (certain water-based liquid) that is no warmer that 37o C.
  Colony forming units (CFU)
  Other Names: Probiotics

SUMMARY:
Primary Objective:

1. To evaluate the safety of orally administered Lactobacillus plantarum strains 299 and 299v, a probiotic, in patients undergoing allogeneic myeloablative HSCT, as measured by incidence of Lactobacillus plantarum bacteremia.

Secondary Objectives:

1. To investigate the feasibility of administering Lactobacillus plantarum 299 and 299v to children and adolescents undergoing HSCT.
2. To describe the overall incidence of bacteremia in HSCT patients who have been administered Lactobacillus plantarum.
3. To describe the overall incidence of acute graft versus host disease (GVHD) in HSCT patients who have been administered Lactobacillus plantarum.

DETAILED DESCRIPTION:
Myeloablative regimens are the backbone of hematopoietic stem cell transplantation (HSCT) and are associated with prolonged periods of cachexia/anorexia, nausea/vomiting, mucositis, and compromised gut integrity (CGI). The toxicities associated with HSCT often lead to prolonged periods of poor oral intake and may result in overt malnutrition. CGI decreases oral tolerance to foods, reduces Quality of Life (QOL) and functional status, delays the transition from the hospital to home setting, and increases the risk of the development of gut-derived infections. Probiotics are nutritional supplements that contain a defined amount of viable microorganisms and upon administration confer a benefit to the host. Clinical trials in adults receiving organ transplants have found probiotics decrease the incidence of infection, the duration of antibiotic use, the incidence of multiorgan failure and systemic inflammation. Children and adolescents undergoing HSCT, experience similar clinical challenges suggesting probiotics may have a therapeutic value in the setting of HSCT. This study is to evaluate the safety and feasibility of administering probiotics to children and adolescents undergoing HSCT.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing myeloablative allogeneic HSCT will be eligible. The source of stem cells can be from bone marrow, umbilical cord blood or cytokine mobilized peripheral blood. Donor can be human leukocyte antigen (HLA) matched sibling or parent, a related donor mismatched for a single HLA locus (class I or II), unrelated marrow or peripheral blood stem cell donor, or unrelated cord blood at least 4/6 antigen match (Class 1 or II).
* Patients of either gender and between 2 and 17.99 years of age
* Patients receiving any type of GVHD prophylaxis are eligible.

Exclusion Criteria:

* Patients who have self-prescribed probiotics within 3 months of starting the conditioning regimen for stem cell transplant (consumption of yogurt products is allowed).
* Patients with known allergy to oats.
* Patients who have had any type of gut damage within the past three months; such as, previous bowel perforations; previous episode of Grade 4 neutropenic colitis or typhlitis.
* Patients with inflammatory bowel syndrome, short small bowel syndrome, Crohns Disease, Ulcerative Colitis, and patients with a history of bowel resections.
* Patients who have undergone a previous allogeneic HSCT.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2010-02; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Neider, MD, Principal Investigator — Johns Hopkins All Children's Hospital; Monica Bhatia, MD, Principal Investigator — Columbia University; Elena J Ladas, PhD, RD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Nemours Children's Clinic, Jacksonville, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Columbia Universtiy Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Lactobacillus Plantarum: There is a single intervention arm in this study. Target accrual for the intervention is 30 subjects. Subjects receive supplementation with Lactobacillus plantarum strains 299 and 299v.
  Lactobacillus plantarum strains 299 and 299v: Patients will receive a daily dose of Lactobacillus plantarum: 1 x10^8 CFU/kg/day. This supplement will be supplied in sachets of powder and will be mixed in water (certain water-based liquid) that is no warmer that 37o C.
  Colony forming units (CFU)
Period: Overall Study
Arm/Group | Lactobacillus Plantarum
Started | 31
Completed | 30
Not Completed | 1
Not completed — < 50% adherence to probiotic | 1

BASELINE CHARACTERISTICS:
Groups:
- Lactobacillus Plantarum: There is a single intervention arm in this study. Target accrual for the intervention is 30 subjects. Subjects receive supplementation with Lactobacillus plantarum strains 299 and 299v.
  Lactobacillus plantarum strains 299 and 299v: Patients will receive a daily dose of Lactobacillus plantarum: 1 x10^8 CFU/kg/day. This supplement will be supplied in sachets of powder and will be mixed in water (certain water-based liquid) that is no warmer that 37o C.
Arm/Group | Lactobacillus Plantarum
Number analyzed (Participants) | 31
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.8 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Lactobacillus Plantarum Bacteremia Infections
Time Frame: 36 days (day -7 to +28 of HSCT)
Population: Children and adolescents undergoing hematopoietic stem cell transplantation (HSCT)
Measure: Number (95% Confidence Interval); unit: Number of infections
Arm/Group | Lactobacillus Plantarum
Number analyzed (Participants) | 30
Number of infections | 0 [0 to 12]

2. Secondary Outcome: Adherence With the Prescribed Dose, Measured as the Percentage of Prescribed Probiotic Doses
Description: To determine the feasibility of administration of L. plantarum 299 and 299v. The treatment is considered feasible for a patient if he/she received at least 50% of the probiotic dose (>= 11 days of treatment).
Time Frame: 22 days (day -7 to +14 of HSCT)
Measure: Median (Full Range); unit: percentage of prescribed doses
Arm/Group | Lactobacillus Plantarum
Number analyzed (Participants) | 30
percentage of prescribed doses | 97 [50 to 100]

3. Secondary Outcome: Number of Non-lactobacillus Infections
Description: To determine incidence of bacteremia in HSCT patients who have been administered lactobacillus plantarum.
Time Frame: 36 days (day -7 to +28 of HSCT)
Measure: Number; unit: Number of non-lactobacillus infections
Arm/Group | Lactobacillus Plantarum
Number analyzed (Participants) | 30
Number of non-lactobacillus infections | 6

4. Secondary Outcome: Number of Acute Graft Versus Host Disease (GVHD) Events in HSCT Patients Who Have Been Administered Lactobacillus Plantarum
Time Frame: Up to Day +100 of HSCT
Measure: Number; unit: Number of GVHD events
Arm/Group | Lactobacillus Plantarum
Number analyzed (Participants) | 30
Number of GVHD events | 9

ADVERSE EVENTS:
Time Frame: Adverse event data were collected and reported up to Day +100
Arm/Group | Lactobacillus Plantarum
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes